CLINICAL TRIAL: NCT06567886
Title: At Home Morning Bright Light Treatment for Chronic Nociplastic Pain
Brief Title: Fibromyalgia Sleep A to ZZZ Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Helen Burgess, Professor of Psychiatry, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00240590; 1R01NR021025-01 (NIH)
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
Keywords: Sleep timing stabilization; Morning light therapy
MeSH Terms: conditions — Fibromyalgia | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Light Therapy (Experimental): All participants will be asked to attend 8 virtual visits over 5 months.
  Participants randomized to the morning light therapy group are asked to wear the glasses for 1 hour per day. The timing of each person's therapy is tailored to their average wake up time during a baseline period. The treatment period is 4 weeks long.
  Interventions: Device: Light Therapy
- Sleep Stabilization (Experimental): All participants will be asked to attend 8 virtual visits over 5 months. Participants randomized to the sleep stabilization arm are asked to follow a fixed sleep schedule tailored to their sleep during a baseline period. The treatment period is 4 weeks.
  Interventions: Behavioral: Sleep Stabilization
- Control Group, treatment as usual (No Intervention): Participants will be asked to sleep as per usual.

INTERVENTIONS:
Device: Light Therapy — Participants will self-administer the daily light therapy within a few minutes of their assigned wake up time for one hour.
  Researchers will provide a light log to note light on/off times, any interruptions to light therapy, and primary activity during light therapy.
  Other Names: Re-Timer
  Arms: Light Therapy
Behavioral: Sleep Stabilization — All participants will be asked to follow a fixed sleep schedule.
  Arms: Sleep Stabilization

SUMMARY:
This research study is testing whether changes in sleep timing and morning light therapy may have an impact on symptoms related to fibromyalgia.

DETAILED DESCRIPTION:
This study will test a consumer health light therapy device (Re-Timer)

ELIGIBILITY:
Inclusion Criteria:

1. Meets 2016 revised diagnostic criteria for fibromyalgia (FM)
2. Has access to video conferencing (including web cameras and audio) and a private space for the remote study visits.

Exclusion Criteria:

1. Significant chronic disease
2. Severe hearing or memory problems
3. Pending medical leave applications at workplace
4. Current pregnancy, breastfeeding, or actively trying to get pregnant
5. Night work or travel outside the eastern time zone within 1 month of the study
6. Other research participation
7. Frequent number of special events during study period (weddings, concerts, exams, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire-Revised (FIQR) score | baseline (Visit 3, day 8) to post-treatment (Visit 7, approximately day 36).
  The FIQR is 21 questions. Each question has 11 boxes similar to a visual analog scale. Questions include the difficulty associated with various physical activities and the severity of symptoms. The score for the questions is on a scale from 0 - 100, where lower scores represented better functional status.

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) score | baseline (Visit 3, day 8) to post-treatment (Visit 7, approximately day 36).
  The BPI consists of 11 questions and assesses for the presence of pain, pain intensity (i.e., worst, least, average, current) and functional interference from pain. A higher score indicates more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Afton Hassett, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be transmitted to and stored at the NHLBI National Sleep Research Resource (NSRR) data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From study completion and up to 7 years following publication.
Access Criteria: Members of the scientific community who would like a copy of the final data sets (i.e., data sets underlying any publication) from this study can request a copy by contacting the principal investigators and/or NSRR.
URL: https://sleepdata.org/

REFERENCES:
- [Derived] Burgess HJ, Rodgers AA, McNeil KA, Mott J, Fejer A, Dereski T, Rizvydeen M, Sibille KT, Kim HM, Cofield C, Burns JW, Shaikh S, Hassett AL. At-Home Morning Bright Light Treatment for Chronic Nociplastic Pain: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2025 Oct 13;14:e75060. doi: 10.2196/75060. PMID 40880266